CLINICAL TRIAL: NCT05395598
Title: Predicting Moderate Thoracic Aortic Aneurysm Evolution: a Longitudinal Study of Systemic Factors in Patients Free of Connective Tissue Disease. .
Brief Title: Incidence of Major Complication in Case of Thoracic Aortic Aneurysm
Acronym: MOTAAR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Santelys Association (Other); Région Nord-Pas de Calais, France (Other); Association de Cardiologie Nord-Pas de Calais (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021_0151; 2022-A00439-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Thoracic Aortic Aneurysm
Keywords: Thoracic aortic aneurysm; Incidence; nocturnal hypertension; Sleep apnea
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thoracic aneurysm is a silent disease with a potential mid-term high risk of death or major complications. Few data are available on the real incidence of major complications in case of small and moderate thoracic aneurysm. Different factors are supposed to increase the risk of aortic enlargement as high blood pressure and sleep disorder breathing. The modality of imaging and clinical follow-up are well defined. In this prospective observational study, the aim to assess the incidence of of major complications during follow-up in a population of patients with a small or moderate thoracic aneurysm. The study will also try to identify systemic factors influencing aneurysm evolution.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of an aortic root aneurysm > 40 mm
* Agreement to participate to a longitudinal study and available for a 5 years follow-up

Exclusion Criteria:

* Presence of comorbidities or pathology with a prognosis of less than 1 year
* Personal or family history of genetically documented elastic tissue disease or patient meeting the GAND clinical criteria suggestive of Marfan disease
* High-grade mitra-aortic valve disease, even if asymptomatic
* Unbalanced hypertension ≥ 180/110 mmHg
* Aneurysm (regardless of thoracic or abdominal location) ≥ 50 mm
* Aneurysm (regardless of thoracic or abdominal location) with documented progression of more than 5 mm over one year
* History of aortic surgery or endovascular intervention and history of type B aortic dissection of medical treatment
* Renal insufficiency on dialysis, or GFR< 30 ml/mn (CKD-EPI)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate thoracic aortic aneurysms for primary prevention
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2031-04-18 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence within 5 years of inclusion of a major aortic even | during the 5 years after inclusion
  This composite end point is defined as the occurrence of:
  * Aneurysm-related death
  * Emergency surgery for threatened aortic rupture or aortic dissection
  * Scheduled surgery for aneurysmal dilatation of more than 5 mm over 1 year
  * Aneurysm progression exceeding 55 mm in diameter
  * Root surgery for management of symptomatic aortic valve disease (insufficiency or narrowing) of high grade defined by tight aortic narrowing (V Max≥4 m/s, mean gradient ≥40mmHg, and area ≤1cm² or severe aortic insufficiency (regurgitated volume≥60 ml, shortening fraction≥ 50%.

SECONDARY OUTCOMES:
Number of Participants with controlled blood pressure defined by ambulatory blood pressure measurement | during the 2 years after inclusion
  The blood pressure measurement (averaged over 24 h)<130/80 mmHg and nocturnal blood pressure ≤120/70 mmHg
Presence of sleep disorders defined by an 'Apnea Hypopnea Index and/or an Oxygen Desaturation Index | during the 2 years after inclusion
  for Apnea Hypopnea Index = ≥5 events per hour for Oxygen Desaturation Index = ≥5 events per hour
Occurrence during the 5 years after inclusion of a major cardiovascular event | during the 5 years after inclusion
  This composite criterion is defined by the occurrence of death from cardiovascular causes, myocardial infarction, stroke (ischemic or hemorrhagic), or hospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DELSART, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU Lille, Lille, Please Choose..., France